CLINICAL TRIAL: NCT06249087
Title: A Randomized Controlled Trial to Explore Effect of Multifunctional Nutrition Tube on Social Condition and Experience in Cerebralvascular Accident
Brief Title: Multifunctional Nutrition Tube on Social Condition and Experience in Cerebralvascular Accident
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zeng Changhao (Other)
Responsible Party: Sponsor-Investigator, Zeng Changhao, Research Director, People's Hospital of Zhengzhou University
Organization: People's Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IOE-XINLI+TIYAN
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the observation group (Experimental): Assigned randomly before the treatment, all patients were provided with comprehensive rehabilitation therapy as follows:
  Basic treatment, including corresponding control of risk factors and education on healthy lifestyles.
  Swallowing training, including lemon ice stimulation, empty swallowing training, and pronunciation training.
  Pulmonary function training, including standing training, cough training, and diaphragm muscle training.
  The observation group was given enteral nutritional support with Intermittent Oro-esophageal Tube according to the following procedure. The feeding content was formulated by the nutritionists based on the condition and relevant guidelines to reach the energy demand as 20-25 kcal/kg/day and protein supplementation of 1.2-2.0 g/kg/day for both two groups
  Interventions: Behavioral: comprehensive rehabilitation therapy; Device: Intermittent Oro-esophageal Tube Feeding
- the control group (Active Comparator): Assigned randomly before the treatment, all patients were provided with comprehensive rehabilitation therapy as follows:
  Basic treatment, including corresponding control of risk factors and education on healthy lifestyles.
  Swallowing training, including lemon ice stimulation, empty swallowing training, and pronunciation training.
  Pulmonary function training, including standing training, cough training, and diaphragm muscle training.
  Besides, the control group was given enteral nutritional support with Nasogastric Tube according to the relevant guidelines. Within 4 hours after admission, the placement of the feeding tube was conducted by professional medical staffs and after intubation, the tube was secured to the cheek with medical tape. The feeding was conducted once every 3-4 hours, with 200-300ml each time. The total feeding volume was determined based on daily requirements.
  Interventions: Behavioral: comprehensive rehabilitation therapy; Device: Nasogastric Tube Feeding

INTERVENTIONS:
Behavioral: comprehensive rehabilitation therapy — Basic treatment, including corresponding control of risk factors and education on healthy lifestyles.
  Swallowing training, including lemon ice stimulation, empty swallowing training, and pronunciation training.
  Pulmonary function training, including standing training, cough training, and diaphragm muscle training.
Device: Intermittent Oro-esophageal Tube Feeding — The observation group was given enteral nutritional support with Intermittent Oro-esophageal Tube according to the following procedure: Before each feeding, inside and outside of the tube was cleaned with water. During feeding, the patient should maintain a semi-reclining or sitting position with mouth opened, and the tube was inserted slowly and smoothly into the upper part of the esophagus by medical staffs while the appropriate depth of intubation was checked with the calibration markings on the tube wall. The distance from the incisors to the head part of the tube should be between 22-25 cm. However, the specific depth should be evaluated based on patients' feedback and adjusted accordingly. After insertion, the tail part of the tube should be put into a container full of water and the absence of continuous bubbles indicated a successful intubation. Then, the feeding was to be conducted three times per day with 50 ml per minute and 400-600ml for each feeding.
  Arms: the observation group
Device: Nasogastric Tube Feeding — The control group was given enteral nutritional support with Nasogastric Tube Feeding according to the relevant guidelines. Within 4 hours after admission, the placement of the feeding tube was conducted by professional medical staffs and after intubation, the tube was secured to the patient's cheek with medical tape. The feeding was conducted once every 3-4 hours, with 200-300ml each time. The total feeding volume was determined based on daily requirements. The feeding content was formulated by the nutritionists based on the patient's condition and relevant guidelines to reach the energy demand as 20-25 kcal/kg/day and protein supplementation of 1.2-2.0 g/kg/day for both two groups. For patients with limited tube feeding compliance, we made appropriate adjustments to ensure that they were not at risk of severe malnutrition as much as possible.
  Arms: the control group

SUMMARY:
The aim of this clinical trial is to compare the psychological condition and experience of ischemic stroke patients who receive enteral nutrition support through either Intermittent Oro-esophageal Tube or Nasogastric Tube. Patients will be randomly assigned to either an observation group or a control group, with both groups receiving routine rehabilitation treatment. The observation group will receive enteral nutrition support through Intermittent Oro-esophageal Tube, while the control group will receive it through Nasogastric Tube. Researchers will then compare the psychological condition and experience of the two groups.

DETAILED DESCRIPTION:
The study will last 15 days for each participant. The goal of this clinical trial is to compare the differences on Psychological Condition and Experience in ischemic stroke patients using Intermittent Oro-esophageal Tube and Nasogastric Tube. Patients will be randomly divided into an observation group and a control group, all receiving routine rehabilitation treatment. On this basis, the observation group will use Intermittent Oro esophageal Tube for enteral nutrition support, while the control group will use Nasogastric Tube. Researchers will compare Psychological Condition and Experience of two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years.
* Meeting the diagnostic criteria for ischemic stroke .
* Dysphagia confirmed by video fluoroscopic Swallowing Study.
* Clear consciousness.
* Stable vital signs.

Exclusion Criteria:

* Dysphagia that might be caused by other diseases that might cause dysphagia, such as head and neck tumors, traumatic brain injury, etc.
* Complicated with severe liver and kidney failure, tumors, or hematological disorders.
* Simultaneously in need to undergo other therapy that might affect the outcomes of this study.
* Pregnant or nursing females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder 7 | day 1 and day 15
  Generalized Anxiety Disorder-7 is a widely used questionnaire to assess the severity of symptoms related to generalized anxiety disorder. The questionnaire consists of 7 questions, each with different answer options. The respondent needs to select the appropriate answer based on their actual condition and assign a corresponding score. The total score ranges from 0-21, with higher scores indicating more severe symptoms.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 | day 1 and day 15
  The total score of the Patient Health Questionnaire-9 ranges from 0 to 27, with higher scores indicating more severe depression symptoms.
Self-made questionnaire | day 1 and day 15
  By conducting a self-made questionnaire, we can assess patients' feelings of fear, shame, uncertainty, and other emotions related to tube feeding. The scores are then converted to a percentage scale ranging from 0 to 100. In the Likert 5-point scale, higher scores indicate worse and more severe conditions for each question.
The Reintegration to Normal Living Index | day 1 and day 15
  The Reintegration to Normal Living Index is a questionnaire used to assess the extent to which individuals have reintegrated into normal life following a stroke. It includes various domains, including social aspects of reintegration. The total score range for the scale is from 0 to 100, and a higher score indicates better reintegration into normal living. Therefore, in the case of the scale, a higher score is considered more favorable as it reflects a greater degree of reintegration into normal life following a stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Study Director — Site Coordinator of United Medical Group located in Miami
Locations (1):
- Khon Kaen Hos., Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No